CLINICAL TRIAL: NCT01659320
Title: Open Treatment of Minocycline in Geriatric Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1005011034; P30MH085943-04 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-08-07 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Minocycline (Experimental): Open label treatment using minocycline.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 100 mg twice daily for 8 weeks

SUMMARY:
This research study will examine whether elderly depressed patients whose depressive symptoms do not respond satisfactorily to therapy with a mood stabilizer or antidepressant alone gain any benefit from taking minocycline alone or in addition to their antidepressant or mood stabilizer medication. Minocycline is a commonly used antibiotic medication with anti-inflammatory properties. It is hoped that information gained from this study will help the investigators better understand the role of inflammation in depression, and whether decreasing inflammation will lead to improvement in the symptoms of depression and cognitive function.

DETAILED DESCRIPTION:
This research study will examine whether elderly depressed patients whose depressive symptoms do not respond satisfactorily to antidepressant therapy alone gain any benefit from taking minocycline alone or in addition to their antidepressants. Minocycline is a commonly used antibiotic medication with anti-inflammatory properties. It is hoped that information gained from this study will help the investigators better understand the role of inflammation in depression, and whether decreasing inflammation will lead to improvement in the symptoms of depression and cognitive function. Elderly patients with depression who remain symptomatic after at least 6 weeks of treatment with an antidepressant medication reaching a therapeutic dosage will be recruited and receive minocycline augmentation for 8 weeks. They may or may not remain on their antidepressants based on their physicians' clinical recommendation. Response to treatment will be measured weekly during the first four weeks and every other week thereafter using rating scales of depressive symptoms, intellectual functions and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Participants must be 55 years old or older (female patients must be postmenopausal);
2. Diagnosis: Major depression, either unipolar or bipolar without psychotic features (by Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria and assessed on the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID);
3. Severity of depression: 17-item Hamilton Depression Rating Scale(HRSD)>14;
4. Failure to achieve substantial improvement of depressive symptoms (entry HDRS>14) after at least 6 weeks of treatment with a mood stabilizer or an antidepressant (SSRI, SNRI, or TCA) reaching therapeutic dosages (daily dose of at least: fluoxetine 20 mg, sertraline 150 mg, paroxetine 20 mg, citalopram 20 mg, escitalopram 10 mg, venlafaxine 150 mg, duloxetine 60 mg).
5. Fluency in English
6. Capacity to provide informed consent.

Exclusion Criteria:

1. High suicide risk, i.e. intent or plan to attempt suicide in near future;
2. Presence of any current Axis I psychiatric disorder (other than unipolar or bipolar major depression or generalized anxiety disorder) including substance abuse (those with a history of substance abuse must be abstinent for at least 3 months prior to entry);
3. Axis II diagnosis of antisocial personality disorder, schizotypal or severe borderline personality, mental retardation and pervasive developmental disorder (DSM-IV);
4. Dementia of more than mild severity (MMSE < 20);
5. History of psychiatric disorders such as psychotic depression, primary psychotic disorder
6. Acute or severe medical illness, i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry, advanced autoimmune deficiency, or "end stage" chronic obstructive pulmonary disease; or drugs known to cause depression, e.g., reserpine, alpha-methyl-dopa, steroids, sympathomimetics withdrawal;
7. Presence of a significant neurological disease such as Parkinson's disease, primary or secondary seizure disorders, intracranial tumors, severe head trauma; neurodegenerative diseases i.e. Multiple Sclerosis;
8. History of intolerance to minocycline or other tetracyclines; use of concomitant drugs that may provide reason to believe that minocycline is contraindicated;
9. Patients on anticoagulants (except low-dose aspirin); patients on ergot alkaloids
10. Patients on MAOIs;
11. Patients' unwillingness or inability to gradually withdraw all other psychotropic medications (except for the following: Antidepressants, mood stabilizers, and low and stable doses of opiates and non-benzodiazepine hypnotics, e.g. zolpidem (5 or 10 mg), zaleplon (5 or 10 mg).
12. Inability to perform any of the ADLs (MAI: ADL subscale) even with assistance, e.g. walking with a cane is not an exclusion criterion;
13. Inability to speak English;
14. Corrected visual acuity < 20/70;

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George S. Alexopoulos, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Institute of Geriatric Psychiatry, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.13 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Asberg Depression Rating Scale total scores range from 0-60. Higher scores indicate greater severity of depression. Total scores are reported with no subscales. Population: We enrolled 16 subjects but 1 subject withdrew consent before any clinical baseline data could be collected.
  units on a scale
    number analyzed (Participants) | 15
    (all) | 24.67 (4.56)
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — MMSE total scores range from 0-30. Higher scores indicate better memory functioning (no cognitive impairment). Total scores are reported with no subscales. Population: We enrolled 16 subjects but 1 subject withdrew consent before any clinical baseline data could be collected.
  units on a scale
    number analyzed (Participants) | 15
    (all) | 28.13 (1.72)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: A published and widely-used scale for rating depression, the Montgomery Asberg Depression Rating Scale total scores range from 0-60. Higher scores indicate greater severity of depression. Total scores are reported with no subscales.
Time Frame: 8 weeks
Population: Among 13 subjects who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline
Number analyzed (Participants) | 13
units on a scale | 16.62 (7.19)

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Arm/Group | Minocycline
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=16)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No